CLINICAL TRIAL: NCT05546931
Title: Multilevel Mobile Health Program to Improve Rural Hypertension
Brief Title: Mobile Health Program for Rural Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jared W Magnani, MD, MSc, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21120151; R01HL160749 (NIH)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hypertension,Essential; Adherence, Medication; Quality of Life
Keywords: hypertension; adherence; rurality
MeSH Terms: conditions — Essential Hypertension; Medication Adherence; Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel-arm, randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A smartphone-based, interactive coaching application designed to enhance adherence to home-based blood pressure monitoring, provided guidance on blood pressure management, patient-facing education, and assistance with modifying behaviors associated with poor blood pressure control; connected to a wireless blood pressure cuff for accurate blood pressure measurement and automated storage on a digital platform. All participants in the experimental arm receive a smartphone for the 6-month intervention duration and the home-based blood pressure cuff.
  Interventions: Behavioral: Coaching application; Behavioral: Home-based blood pressure monitoring
- Enhanced usual care (Active Comparator): WebMD, a smartphone-based tool for learning about blood pressure and other health conditions. Enhanced usual care participants receive a wireless blood pressure cuff for accurate blood pressure measurement and automated storage on a digital platform. All participants in the experimental arm receive a smartphone for the 6-month intervention duration and the home-based blood pressure cuff.
  Interventions: Other: WebMD; Behavioral: Home-based blood pressure monitoring

INTERVENTIONS:
Behavioral: Coaching application — A digital application for providing education and support for home-based blood pressure monitoring.
  Arms: Intervention
Other: WebMD — Smartphone-based application for health education and/or monitoring.
  Arms: Enhanced usual care
Behavioral: Home-based blood pressure monitoring — Device for measuring blood pressure at home with blue tooth connectivity for automated collection.

SUMMARY:
Hypertension (HTN) is the leading modifiable cause of cardiovascular disease. Rural individuals experience challenges of the rural health divide: geographic distance from providers, social isolation, limited social resources, and high rates of low health literacy. This study evaluates a home-based blood pressure monitoring (HBPM) program that provides longitudinal health education, empathic guidance, monitoring, and adaptable patient-centered coaching to rural individuals. Participants in this study will be randomized to receive (1) HBPM with the intervention; or (2) the control, consisting of HBPM and a smartphone with a general health application (WebMD).

DETAILED DESCRIPTION:
Hypertension (HTN) has increasing prevalence, is the leading cause of cardiovascular morbidity and mortality, and contributes significantly to health care utilization and costs. Social determinants of health (SDOH) exacerbate patients' access to therapies, adherence, and health outcomes. A robust literature demonstrates the effects of income, education, health literacy, and social resources on access to HTN treatment; medication adherence; and short- and long-term likelihood of clinical adversity. In the U.S., geographic obstacles to care further complicate HTN treatment and outcomes for rural individuals. This single-center, parallel group randomized clinical trial (RCT) evaluates a home-based blood pressure monitoring (HBPM) and cardiovascular mobile health platform in rural individuals with hypertension (HTN). The intervention uses a virtual coaching platform to provide health education, monitoring, guidance, and adaptable patient-centered coaching to rural individuals. The 6-month intervention provides a personalized curriculum to promote HBPM; medication adherence; HTN education; non-pharmacologic strategies for HTN management; preparation for the clinical encounter; and enhanced problem-solving and engagement for rural individuals. The trial is 12-month duration with visits at baseline, 6, and 12 months. Individuals with poorly controlled HTN (systolic BP 140-199 or diastolic BP 90-119 mm Hg at 2 ambulatory visits) will be randomized to: (1) intervention, the HBPM coaching intervention and HBPM; or (2) control, smartphone with a general health application (WebMD) and HBPM. For both intervention and control, summaries of BP measures are provided to clinicians in order to improve HTN management for rural patients. The primary study outcome is improvement in BP from baseline to 6 months. The secondary study outcomes are comparison of adherence to antihypertensive medications and patient-reported outcomes in the intervention and usual care arms at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. History of uncontrolled hypertension, identified from the electronic health record problem list and an average systolic BP 140-199 or diastolic BP 90-119 mm Hg at 2 ambulatory visits, one of which is within 6 months of study entry
2. Residence in one of 48 counties categorized as rural by the Center for Rural Pennsylvania;
3. English-speaking at level appropriate for informed consent and study participation;
4. No plans to relocate from the area within 12 months of enrollment.

Exclusion Criteria:

1. Heart failure necessitating hospital admission ≤3 months prior to study inclusion;
2. Acute coronary syndrome (defined as at least 2 of the following: chest pain, ischemic electrocardiographic changes, or troponin ≥0.1 ng/mL) ≤3 months prior to study inclusion;
3. Planned major surgery, cardiovascular or non-cardiovascular;
4. Pregnancy or planned pregnancy within 12 months;
5. Presence of non-cardiovascular conditions likely to be fatal within 12 months (e.g., cancer);
6. Inability to comprehend the study protocol, defined by failing 3 times to answer correctly a set of questions during consent;
7. Institutionalized status (e.g., nursing home, incarceration);
8. Inability to operate a smartphone or HBPM device due to sensory or neurocognitive deficit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure from baseline to 6 months | Baseline, 6 months
  Change in home-based systolic and diastolic blood pressure from baseline to 6 months between the intervention and usual care arms.

SECONDARY OUTCOMES:
Adherence to antihypertensive medications | Baseline, 6 months
  Adherence to antihypertensive medication from baseline to 6 months between the intervention and usual care arms using Proportion of Days Covered, ranging from 0 to 100%, where higher values indicate superior medication adherence.
Adherence to antihypertensive medications | Baseline, 12 months
  Adherence to antihypertensive medication from baseline to 12 months between the intervention and usual care arms using Proportion of Days Covered, ranging from 0 to 100%, where higher values indicate superior medication adherence.
Patient-Reported Outcomes | Baseline, 6 months
  Patient-reported outcomes between the intervention and usual care arms at 6 months measured with the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) with distinct assessments of the following: (1) physical function, (2) anxiety, (3) depression, (4) fatigue, (5) sleep, (6) ability to participate in social roles, (7) social role satisfaction, and (8) interference in functioning by pain. Each domain is scored separately, such that scores for each domain range from 4 (lowest score) to 20 (highest score), where higher scores indicate greater impairment.
Patient-Reported Outcomes | Baseline, 12 months
  Patient-reported outcomes between the intervention and usual care arms at 12 months measured with the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) with distinct assessments of the following: (1) physical function, (2) anxiety, (3) depression, (4) fatigue, (5) sleep, (6) ability to participate in social roles, (7) social role satisfaction, and (8) interference in functioning by pain. Each domain is scored separately, such that scores for each domain range from 4 (lowest score) to 20 (highest score), where higher scores indicate greater impairment.
Self-efficacy for managing medications and treatment | Baseline, 6 months
  Patient-reported outcomes between the intervention and usual care arms at 6 months measured with the Patient-Reported Outcomes Measurement Information System Self-efficacy for managing medications and treatment, a 10-item instrument, scored from 10 (minimum) to 40 (maximum), where higher scores indicate superior self-efficacy.
Self-efficacy or managing medications and treatment | Baseline, 12 months
  Patient-reported outcomes between the intervention and usual care arms at 12 months measured with the Patient-Reported Outcomes Measurement Information System Self-efficacy for managing medications and treatment, a 10-item instrument, scored from 10 (minimum) to 40 (maximum), where higher scores indicate superior self-efficacy.
Adherence to home blood pressure monitoring | From enrollment to the end of the intervention phase at 6 months.
  Quantification of home blood pressure monitoring during the 6-month intervention phase, characterized as both a continuous and categorical measure, compared by study arm.

OTHER OUTCOMES:
Change in systolic and diastolic blood pressure from baseline to 6 months, stratified by home-supervised blood pressure at baseline visit. | Baseline, 6 months
  Change in home-based systolic and diastolic blood pressure from baseline to 6 months between the intervention and usual care arms, stratified by home-supervised blood pressure at baseline visit (systolic BP <130 or >=130 mm Hg; diastolic BP <85 or >=85 mm Hg in separate analyses).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will share all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available 12 months following publication of the primary results of this trial.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to the Principal Investigator at magnanij@pittt.edu. To gain access, data requestors will need to sign a data access agreement. Data will be provided directly by the study investigators. Costs associated with producing datasets and analysis will be the responsibility of investigators seeking the data.